CLINICAL TRIAL: NCT00497302
Title: Recovery Housing For Drug Dependent Pregnant Women
Acronym: HOME
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Hendree E. Jones, Adjunct Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA014979 (NIH); R01DA014979 (NIH); DPMCDA
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Drug Addiction
Keywords: cocaine; opiate; pregnancy; post-partum; neonatal abstinence syndrome; contingency management; Reinforcement Based Treatment; women
MeSH Terms: conditions — Substance-Related Disorders; Neonatal Abstinence Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): receives housing based on drug abstinence
  Interventions: Behavioral: RBT
- 2 (Active Comparator): Usual care treatment at the Center for Addiction and Pregnancy
  Interventions: Behavioral: usual care

INTERVENTIONS:
Behavioral: RBT — Contingency management and behavioral counseling including motivational interviewing
  Arms: 1
Behavioral: usual care — receives usual comprehensive care at Center for Addiction and Pregnancy
  Arms: 2

SUMMARY:
For the past several years our research program has developed and tested an intensive outpatient intervention that is based in social learning theory and employs abstinence contingent access to recovery housing as a routine aspect of an intensive day treatment counseling program. The present project proposes to extend this treatment intervention to the special population of pregnant drug using women enrolled at the Center for Addiction and Pregnancy (CAP). We will compare an enhanced treatment that includes abstinence contingent recovery house living plus intensive individual therapy, to standard care at the CAP program. Specific aims of the project are derived from testing a two-group design are described below:

1. To determine whether financially supported abstinence-contingent recovery house placement plus individual counseling in pregnant drug-dependent women improves prenatal outpatient treatment retention.
2. To determine whether financially supported abstinence-contingent recovery house placement plus individual counseling in pregnant drug-dependent women reduces prenatal drug use.
3. To determine whether financially supported abstinence-contingent recovery house placement plus individual counseling results in better maternal and infant clinical birth outcomes (e.g., birth weight, estimated gestational age (EGA) at delivery, medical complications).

ELIGIBILITY:
Inclusion Criteria:

* CAP enrolled
* Age 18 or older
* Evidence of use of opiate and/or cocaine use in the past 30 days
* Assigned to pharmacotherapy free modality
* CAP admission at an estimated gestational age (EGA) <34 weeks

Exclusion criteria:

* Endorses current suicidal ideation
* Any medical disorders requiring extended or future hospitalization
* Meet diagnostic criteria for current DSM-IV alcohol dependence
* Meet diagnostic criteria for a current DSM-IV Axis I thought disorder (i.e. schizophrenia)
* Demonstrate significant cognitive impairment that precludes them from completing the initial assessment battery

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2004-11; Primary Completion 2008-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Treatment retention, drug free urine samples at follow-up and delivery | treatment entry until 12 months post treatment entry

SECONDARY OUTCOMES:
prenatal care compliance, neonatal and birth outcomes | treatment entry until 12 months post treatment entry

CONTACTS AND LOCATIONS:
Overall Officials: Hendree E Jones, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Center for Addiction and Pregnancy Jhons Hopkins Bayview Medical Center, Baltimore, Maryland, United States